CLINICAL TRIAL: NCT06224816
Title: Clinical Trial to Assess the Clinical Impact, Efficacy and Safety of Customized Nasal Masks Designed by 3D Printing During Non-invasive Ventilation in Premature Infants
Brief Title: Clinical Trial for the Evaluation of Customized 3D Printed NIV Nasal Masks in Premature Infants
Acronym: M3DPREMAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: ISCIII (Unknown)
Responsible Party: Principal Investigator, María Teresa Moral Pumarega, Associate Professor of Pediatrics at the Complutense University of Madrid (UCM), Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M3DPREMAT
Record Dates: First submitted 2023-12-20; First posted 2024-01-25 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Premature Lungs
Keywords: Neonatology; Nasal mask; 3D printing; Additive manufacturing; Newborn; Premature; Prematurity; Neonate; Non-Invasive Ventilation (NIV); Oxygen saturation; SolidWorks; 3D scanner; Customized device; Continuous positive airway pressure (CPAP)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Mask (3DM) (Experimental): Custom 3D mask (3DM) application in neonate during 4 hours. Each patient included will be their own control at the same time, receiving each of the different mask models every 4 hours alternately. The study period will be a maximum of 7 days.
  Interventions: Device: Custom 3D mask (3DM) application in neonate; Device: Traditional mask (TM) application in neonate
- Traditional Mask (TM) (Active Comparator): Traditional Mask (TM) application in neonate during 4 hours. Each patient included will be their own control at the same time, receiving each of the different mask models every 4 hours alternately. The study period will be a maximum of 7 days.
  Interventions: Device: Custom 3D mask (3DM) application in neonate; Device: Traditional mask (TM) application in neonate

INTERVENTIONS:
Device: Custom 3D mask (3DM) application in neonate — Premature infants with a birth weight less than 1500 g r first received 3D mask during 4 hour, then crossed over to traditional mask.
Device: Traditional mask (TM) application in neonate — Premature infants with a birth weight less than 1500 g r first received traditional mask during 4 hours, then crossed over to 3D mask.

SUMMARY:
Clinical trial with crossed groups, open, masked for the evaluation of the main outcome. Inclusion of all premature infants with a birth weight less than 1500 g requiring Non-invasive Ventilation (NIV).

Premature will be randomised to start alternatively with MT or 3DM. Each patient included will be their own control at the same time, receiving each of the different mask models every 4 hours alternately. The study period will be a maximum of 7 days.

To compare the time in which preterm maintain SatO2 below 85% with the 3DM versus the traditional mask (TM) in preterm < 1500 g. Other secondary objectives regarding ventilation enhancement will be assessed, such as the number of bradycardias, cardiorespiratory arrest and need for resuscitation in the context of apnea. Also, skin lesions of the nose resulting from the pressure applied by any of the masks (TM or 3DM) and the need for analgesia and/or sedation for pain control or discomfort will be assessed. Parental perception and satisfaction will be assessed.

DETAILED DESCRIPTION:
Improvement and optimization of non-invasive ventilation (NIV) in preterm and low birth weight infants is essential in order to reduce morbidity. By the use of 3D printing design (3DM), these infants would be provided with customized nasal masks, according to their particular anatomical features while on NIV. This would lead to a greater stabilization of the respiratory system, decreased apnea spells, oxygen desaturation and bradycardia, less need for intubation and less skin nose injury, all of which might improve neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newborn prematurity
* Age: less than 30 days of life
* Required respiratory support with non-invasive ventilation (NIV)
* Premature infant has not been on NIV for more than 3 days before being included in the trial.
* Signature of the Informed Consent (IC)

Exclusion Criteria:

* Failure to meet entry criteria
* Cyanotic congenital heart disease diagnosis
* Presence of serious malformations
* Presence of airway malformations

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time in which preterm maintain SatO2 below 85%. | 7 days
  To compare the time in which preterm maintain SatO2 below 85%.in the period of time that customized 3D printed nasal mask (3DM) is used versus traditional nasal mask (TM).

SECONDARY OUTCOMES:
Time in which preterm maintain bradycardias. | 7 days
  To compare the time in which preterm maintain bradycardias - heart rate below 100 beats per minute - that occur in the period of time that customized 3D printed nasal mask (3DM) is used versus traditional nasal mask (TM).
Time in which preterm maintain SatO2 below 75%. | 7 days
  To compare the time in which preterm maintain SatO2 below 75%.in the period of time that customized 3D printed nasal mask (3DM) is used versus traditional nasal mask (TM).
Number of times requiring cardiopulmonary resuscitation | 7 days
  Compare the number of times requiring cardiorespiratory resuscitation with self-inflating bag in the context of apnea pause or severe desaturation in the period of time that customized 3D printed nasal mask (3DM) is used versus traditional nasal mask (TM).
Appearance of cutaneous lesions in nasal region or mucosa | 7 days
  To compare the appearance of cutaneous lesions in the nasal region or nasal mucosa as a consequence of the pressure exerted by any of the masks, indicating the location and degree of the wound in the period of time that customized 3D printed nasal mask (3DM) is used versus traditional nasal mask (TM).
Pain assessment with scoring scale. | 7 days
  To compare the degrees of pain, measured in the neonatal pain scale PIPP-R (Premature Infant Pain Profile-Revised), obtained every 12 hours in the period of time that customized 3D printed nasal mask (3DM) is used versus traditional nasal mask (TM). Regarding the PIPP-R scale, the minimum score is 1 and the maximum is 21. Scores between 1-6 correspond to mild pain, 7-11 moderate pain, and 12-21 severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: María Teresa Moral Pumarega, Principal Investigator — Hospital Universitario 12 de Octubre; Antonio Martín González, Mechanical Engineering, Study Chair — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Ramahi J, Luo H, Fang R, Chou A, Jiang J, Kille T. Development of an Innovative 3D Printed Rigid Bronchoscopy Training Model. Ann Otol Rhinol Laryngol. 2016 Dec;125(12):965-969. doi: 10.1177/0003489416667742. Epub 2016 Sep 7. PMID 27605436
- [Background] Zheng J, He H, Kuang W, Yuan W. Presurgical nasoalveolar molding with 3D printing for a patient with unilateral cleft lip, alveolus, and palate. Am J Orthod Dentofacial Orthop. 2019 Sep;156(3):412-419. doi: 10.1016/j.ajodo.2018.04.031. PMID 31474271
- [Background] Hadeed K, Dulac Y, Acar P. Three-dimensional printing of a complex CHD to plan surgical repair. Cardiol Young. 2016 Oct;26(7):1432-4. doi: 10.1017/S1047951116000755. Epub 2016 Jun 20. PMID 27321706
- [Background] Xu JJ, Luo YJ, Wang JH, Xu WZ, Shi Z, Fu JZ, Shu Q. Patient-specific three-dimensional printed heart models benefit preoperative planning for complex congenital heart disease. World J Pediatr. 2019 Jun;15(3):246-254. doi: 10.1007/s12519-019-00228-4. Epub 2019 Feb 22. PMID 30796731
- [Background] Zhao H, Lin G, Seong YH, Shi J, Xu J, Huang W. Anthropometric research of congenital auricular deformities for newborns. J Matern Fetal Neonatal Med. 2019 Apr;32(7):1176-1183. doi: 10.1080/14767058.2017.1402877. Epub 2017 Dec 8. PMID 29219007
- [Background] Minocchieri S, Burren JM, Bachmann MA, Stern G, Wildhaber J, Buob S, Schindel R, Kraemer R, Frey UP, Nelle M. Development of the premature infant nose throat-model (PrINT-Model): an upper airway replica of a premature neonate for the study of aerosol delivery. Pediatr Res. 2008 Aug;64(2):141-6. doi: 10.1203/PDR.0b013e318175dcfa. PMID 18391845
- [Background] Saugstad OD, Aune D. Optimal oxygenation of extremely low birth weight infants: a meta-analysis and systematic review of the oxygen saturation target studies. Neonatology. 2014;105(1):55-63. doi: 10.1159/000356561. Epub 2013 Nov 15. PMID 24247112
- [Background] Stenson BJ. Oxygen targets for preterm infants. Neonatology. 2013;103(4):341-5. doi: 10.1159/000349936. Epub 2013 May 31. PMID 23736013
- [Background] Bose CL, Dammann CE, Laughon MM. Bronchopulmonary dysplasia and inflammatory biomarkers in the premature neonate. Arch Dis Child Fetal Neonatal Ed. 2008 Nov;93(6):F455-61. doi: 10.1136/adc.2007.121327. Epub 2008 Aug 1. PMID 18676410
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433
- [Background] Sweet DG, Carnielli VP, Greisen G, Hallman M, Klebermass-Schrehof K, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome: 2022 Update. Neonatology. 2023;120(1):3-23. doi: 10.1159/000528914. Epub 2023 Feb 15. PMID 36863329
- [Background] Roh S, Parekh DP, Bharti B, Stoyanov SD, Velev OD. 3D Printing by Multiphase Silicone/Water Capillary Inks. Adv Mater. 2017 Aug;29(30). doi: 10.1002/adma.201701554. Epub 2017 Jun 7. PMID 28590510
- [Background] Hinton TJ, Hudson A, Pusch K, Lee A, Feinberg AW. 3D Printing PDMS Elastomer in a Hydrophilic Support Bath via Freeform Reversible Embedding. ACS Biomater Sci Eng. 2016 Oct 10;2(10):1781-1786. doi: 10.1021/acsbiomaterials.6b00170. Epub 2016 May 4. PMID 27747289
- [Background] Bhattacharjee N, Parra-Cabrera C, Kim YT, Kuo AP, Folch A. Desktop-Stereolithography 3D-Printing of a Poly(dimethylsiloxane)-Based Material with Sylgard-184 Properties. Adv Mater. 2018 May;30(22):e1800001. doi: 10.1002/adma.201800001. Epub 2018 Apr 14. PMID 29656459
- [Background] Clarke A, Yeomans E, Elsayed K, Medhurst A, Berger P, Skuza E, Tan K. A randomised crossover trial of clinical algorithm for oxygen saturation targeting in preterm infants with frequent desaturation episodes. Neonatology. 2015;107(2):130-6. doi: 10.1159/000368295. Epub 2014 Dec 12. PMID 25531240
- [Background] Duong K, Glover J, Perry AC, Olmstead D, Ungrin M, Colarusso P, MacLean JE, Martin AR. Feasibility of three-dimensional facial imaging and printing for producing customised nasal masks for continuous positive airway pressure. ERJ Open Res. 2021 Feb 1;7(1):00632-2020. doi: 10.1183/23120541.00632-2020. eCollection 2021 Jan. PMID 33569497
- [Background] Kamath AA, Kamath MJ, Ekici S, Stans AS, Colby CE, Matsumoto JM, Wylam ME. Workflow to develop 3D designed personalized neonatal CPAP masks using iPhone structured light facial scanning. 3D Print Med. 2022 Aug 1;8(1):23. doi: 10.1186/s41205-022-00155-7. PMID 35913689